CLINICAL TRIAL: NCT00164411
Title: Pneumococcal Conjugate Vaccine (Prevnar; Wyeth) With Pneumococcal Polysaccharide Vaccine (23-valent) and Tetanus/Diphtheria Vaccine
Brief Title: Pneumococcal Conjugate Vaccine With Pneumococcal Polysaccharide Vaccine and Tetanus/Diphtheria Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Emory University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NIP-3669
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Pneumococcal Infections
Keywords: Diptheria-Tetanus vaccine; Pneumococcal vaccine; Adverse events following vaccination; Immunization; Immunogenicity
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine; 23-valent pneumococcal capsular polysaccharide vaccine

INTERVENTIONS:
Biological: Tetanus-diphtheria toxoids (Td)
Biological: 7-valent pneumococcal conjugate vaccine
Biological: 23-valent polysaccharide vaccine

SUMMARY:
The purpose of this study is to learn whether or not giving a tetanus/diphtheria vaccination ("tetanus shot") before giving pneumococcal vaccine makes the pneumococcal vaccine more effective without causing too many side effects.

DETAILED DESCRIPTION:
The only vaccine licensed in the United States for protecting adults against pneumococcal disease (PPV23) protects against invasive disease in observational studies but has generally been poorly effective against pneumonia or all-cause mortality in randomized clinical trials. Another vaccine containing seven polysaccharide antigens conjugated to diphtheria toxoid (PCV7) is licensed for children and under investigation in adults.

In this pilot study, we are comparing the safety and immunogenicity of three immunization schedules in adults:

* Td vaccine, 2-week interval, PCV7, 4-month interval, PPV23
* PCV7, 4-month interval, PPV23
* PPV23

We aim to:

* compare the safety profiles of pneumococcal vaccines given on each of the three schedules
* compare serotype-specific ELISA antibody response to pneumococcal antigens given on each of the three schedules
* compare functional serotype-specific antibody responses to pneumococcal antigens given on each of the three schedules
* study the influence of diphtheria antibody levels at the time of pneumococcal conjugate vaccine administration on the magnitude of the immune response to pneumococcal antigens

ELIGIBILITY:
Exclusion Criteria:

* Participation in any other investigational clinical trials except purely observational studies within 4 weeks prior to study start
* Any vaccination within 2 weeks prior to first study vaccine
* Evidence of systemic or local infection within one week prior to first study vaccine
* HIV infection
* Renal failure
* Receipt of a pneumococcal or Td vaccine within 5 years
* Current receipt of therapy for neoplastic disease
* Current receipt of immunosuppressive therapy
* Terminal illness withlife expectancy less than 3 months

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2004-01; Study Completion 2005-03

PRIMARY OUTCOMES:
ELISA for S. pneumoniae antibody 2 months after receiving PPV23
Functional S. pneumoniae antibody 2 months after receiving PPV23

SECONDARY OUTCOMES:
Incidence of adverse events following vaccination from entry to 2 months after receiving last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Harry L Keyserling, MD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States